CLINICAL TRIAL: NCT04073355
Title: Smart Walk 50+: Feasibility of a Smartphone-delivered Physical Activity Program for African American Women 50 Years and Older
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Rodney P Joseph, Assistant Professor, Arizona State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00010333
Record Dates: First submitted 2019-08-26; First posted 2019-08-29 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Physical Activity
Keywords: exercise; African American women; mHealth; eHealth; smartphone
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Activity (Experimental): Smartphone-delivered physical activity intervention
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — Smartphone-delivered physical activity intervention

SUMMARY:
The purpose of this study is to establish the acceptability and feasibility of a culturally relevant, theory-based smartphone-delivered physical activity intervention among African American women aged 50-65 years.

DETAILED DESCRIPTION:
This study will establish the acceptability and feasibility of a culturally relevant, theory-based smartphone-delivered physical activity intervention among African American women aged 50-65 years. To accomplish this, we will deliver our previously developed Smart Walk physical activity intervention, originally developed for African American women aged 24-50 years old, to 20 sedentary and obese African American women aged 50 to 65. We will collect data on the acceptability and feasibility of the intervention, as well as areas of intervention refinement to enhance the social, cultural, and behavioral relevance of the intervention for women in this age group.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported African American female
* Between the ages of 50 to 65
* Insufficiently Active (less than or equal to 60 mins of moderate-to-vigorous physical activity/week measured by Exercise Vital Sign Questionnaire)
* BMI > 30
* English speaking and reading

Exclusion Criteria:

* Plans to relocate out of Phoenix area in next 6 months
* Endorsing an item on the PAR-Q, unless a doctor's note for study participation in provided
* Self-reported participation in another diet or weight loss study
* Non-English reading and speaking
* Pregnant or planning to become pregnant in the next 6 months

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 20 (Actual)
Dates: Start 2019-08-10 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Acceptability and Feasibility: Treatment Acceptance | 4 months
  Treatment acceptance will be assessed via a post-intervention treatment acceptance survey and qualitative data from a post-intervention focus group.
Acceptability and Feasibility: Number of participants who complete 4-month follow-up assessments | 4 months
  Number of participants who complete 4-month follow-up assessment

SECONDARY OUTCOMES:
Changes in Objectively-measured Physical Activity | 4 months
  Pre-post intervention changes in physical activity measured by accelerometers
Changes in self-reported Physical Activity | 4 months
  Pre-post intervention changes in self-reported physical activity as measured by the REGICOR questionnaire
Changes in Exercise Self-efficacy | 4-months
  Pre-post intervention changes in exercise self-efficacy. Assessed by the Exercise Confidence Survey (Sallis, 1988).
Changes in Outcome Expectations for Exercise | 4-months
  Pre-post intervention changes in outcome expectations for exercise; assessed by the Outcome Expectation Scale for Exercise (Resnick, 2000
Changes in Physical Activity Self-regulation | 4-months
  Pre-post intervention changes in self-regulation for physical activity; assessed by the Self-Regulation Scale from the Health Beliefs Survey (Anderson, 2010)
Changes in Social Support for Exercise | 4-months
  Pre-post intervention changes in social support for exercise; assessed by the Social Support for Exercise Survey (Sallis,1987)
Changes in Physical Activity Knowledge | 4-months
  Pre-post intervention changes in knowledge of the national physical activity guidelines; assessed by a 6 item scale developed by study authors

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joseph RP, Ainsworth BE, Hollingshead K, Todd M, Keller C. Results of a Culturally Tailored Smartphone-Delivered Physical Activity Intervention Among Midlife African American Women: Feasibility Trial. JMIR Mhealth Uhealth. 2021 Apr 22;9(4):e27383. doi: 10.2196/27383. PMID 33885368